CLINICAL TRIAL: NCT00623051
Title: Evaluation of the Extension at Community Level of Safe Male Circumcision (ANRS 12126 ORANGE FARM 2)
Acronym: ORANGE FARM 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Responsible Party: Sponsor
Organization: ANRS, Emerging Infectious Diseases (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ANRS 12126 ORANGE FARM 2
Record Dates: First submitted 2008-02-11; First posted 2008-02-25 (Estimated); Last update posted 2013-07-17 (Estimated); Status verified 2013-07

CONDITIONS: HIV Infections
Keywords: male circumcision; HIV; sexual behavior; HIV prevention; HIV Seronegativity
MeSH Terms: conditions — HIV Infections; Sexual Behavior | interventions — Circumcision, Male

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Male circumcision by experimented doctor or nurse
  Interventions: Procedure: Male Circumcision

INTERVENTIONS:
Procedure: Male Circumcision

SUMMARY:
This study is aimed at demonstrating whether or not Male Circumcision can be used as an effective public health prevention tool that will have an impact on HIV prevalence in the South African population.

DETAILED DESCRIPTION:
A randomized, controlled trial (ANRS 1265) conducted in Orange Farm (South Africa) has demonstrated that male circumcision (MC) can reduce the risk of HIV acquisition by more than 50% among young men. This result has been confirmed by two similar studies conducted in Uganda and in Kenya.

Giving these findings, the next logical step is to demonstrate whether or not MC can be used as an effective public health prevention tool that will have an impact on HIV in populations as well as among individuals.

This research study aims to establish a MC intervention in the community where the first randomized controlled trial of the impact of MC on men's risk of acquiring HIV infection was carried out in order to evaluate its impact on:

1. knowledge, attitudes and practice regarding MC
2. existing means of prevention (sexual behavior change, condom use, STI treatment-seeking behavior and VCT (voluntary counseling and testing) attendance)
3. the spread of HIV and HSV-2

This research will be carried out over a period of 60 months and will have three major components: (1) the delivery of the intervention, (2) quantitative studies (cross-sectional surveys), and (3) qualitative studies.

ELIGIBILITY:
Inclusion Criteria:

* being uncircumcised
* living in Orange Farm (South Africa) for more than 3 months
* agreeing to follow the instructions given by doctors, nurses and/or staff, and in particular to abstain from sex for 6-weeks after being circumcised
* having understood and sign a consent form written in their own language
* for those younger than 18 years of age having a written authorization from one parent or guardian and having signed an assent form.

Exclusion Criteria:

* subjects with contraindications for male circumcision
* allergy to anesthesia
* hemophilia or bleeding disorders
* genital ulceration or other symptoms of sexually transmitted infections
* signs of infections or AIDS
* abnormal genital anatomy
* history of diabetes

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 27000 (Actual)
Dates: Start 2008-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
HIV prevalence in population | at the end of the study

SECONDARY OUTCOMES:
Sexual behavior, HSV-2 prevalence, circumcision prevalence, knowledge regarding HIV, AIDS and male circumcision | at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Bertran Auvert, MD, PhD, Principal Investigator — University of Versailles, INSERM U687, France; David Lewis, MD, Principal Investigator — NICD, Johannesburg; Mohamed Haffejee, MD, Principal Investigator — Wits Medical School, Urology Department, Johannesburg
Locations (1):
- Male Circumcision Centre, Orange Farm, Johannesburg, South Africa

REFERENCES:
- See also: Related Info — http://www.anrs.fr